CLINICAL TRIAL: NCT06226740
Title: Evaluation of the Effects of Different Obturation Techniques on Postoperative Pain and Radiographic Healing Non Surgical Endodontic Retreatment in Single Visit in Teeth With Single Root Canals and Apical Periodontitis
Brief Title: Effectiveness of Different Obturation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Merve Işık, Assistant Professor Dr, Abant Izzet Baysal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-DHF-MI-01
Record Dates: First submitted 2023-12-04; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Apical Periodontitis; Postoperative Pain; Endodontically Treated Teeth
Keywords: warm vertical compaction; single visit; postoperative pain; non-surgical endodontic retreatment; cold lateral compaction; numeric rating scale
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold Lateral Compaction (Control group) (Experimental): After the root canal preparation was completed, the working length was checked with the master cone and periapical radiography. The master cone was then covered with root canal sealer and placed in the root canal. Then, a gap was created for the .02 angled lateral cones using #30, 25 and 20 finger spreader. The obturation process continued until the spreader went 2 mm beyond the level of the canal orifice. Next, a hot excavator removed the coronal gutta-percha 1 mm below the canal orifice.
  Interventions: Other: Single Visit Non Surgical Root Canal Treatment Protocol
- Warm Vertical Compaction (Experimental): After the root canal preparation was completed, the working length was checked with the master cone and periapical radiography. Root canal sealer was applied to the root canal walls using a master cone. HeatPlugger connected to the down-pack unit of the obturation system was adjusted to be 4 mm shorter than the working length. The master cone was cut 1 mm shorter than the working length with a heated plugger and applied to the root canal. Then, the heated plugger was advanced in the apical direction, and the apical region was obturated. Obturation was completed in 2 stages with gutta-percha in the gutta-percha cartridge connected to the remaining root canal cavity back-fill unit and heated to 200 °C. Heated gutta-percha was vertically condensed with HeatPlugger to 1 in the first stage and 2 in the second. The root canal obturation was completed by removing the gutta-percha 1 mm below the canal orifice.
  Interventions: Other: Single Visit Non Surgical Root Canal Treatment Protocol
- Gutta Core (Experimental): After the root canal preparation was completed, the working length was controlled with the master cone and periapical radiography. Root canal sealer was applied to the root canal walls using a master cone. Root canal obturation was completed with heated gutta-percha according to the manufacturer's instructions. The heated gutta-percha was slowly inserted into the canal up to the working length. After cutting the handle of the obturators at the level of the canal orifice with a hot excavator, it was condensed into the canal using a gutta-percha plugger. The coronal gutta-percha was removed 1 mm below the canal orifice using a hot excavator.
  Interventions: Other: Single Visit Non Surgical Root Canal Treatment Protocol

INTERVENTIONS:
Other: Single Visit Non Surgical Root Canal Treatment Protocol — The current study aimed to compare the effects of different obturation techniques on postoperative pain level and radiographic healing in non-surgical endodontic treatment applied in a single visit in teeth with single root canal and apical periodontitis.

SUMMARY:
Aim: Evaluation of the effect of different obturation techniques on postoperative pain level and radiographic healing on non-surgical endodontic retreatment (NSER) applied in a single visit in teeth with single root canal and apical periodontitis (AP).

Materials and Methods: 63 teeth with single-root canal and AP from 50 systemically healthy patients (mean age 34.19±9.75 years; 27 women, 23 men) were included in the study. Residual root canal filling materials were removed with retreatment files. All teeth were prepared using rotary files . The teeth were randomly divided into three groups according to the obturation technique; cold lateral compaction (CLC), continuous wave compaction (CWC), and gutta-core (TGC). Restorations are completed using direct composite resin in the same visit. In all cases, pain status were evaluated using the Numerical Pain Rating Scale (NRS) at preoperative, postoperative, 3rd hour, 24th hour, 48th hour, and 7th day. Periapical index (PAI) scores were recorded on preoperative and postoperative 6-month on the periapical radiographs for cases. Data were analyzed as statistically. Significance level was determined as p < 0.05.

DETAILED DESCRIPTION:
All procedures were performed by a endodontist (XX) only in patients who met the inclusion criteria. All patients were informed about the risks of the study and alternative treatment options before participating. Anaesthesia was achieved with 4% articaine hydrochloride containing 1:100,000 adrenalin. None of the patients required additional anaesthesia. After rubber dam isolation, previous caries and restorations were removed with high and low speed sterile burs under water cooling. The previous root canal obturation of all teeth included in the study was removed with a similar treatment protocol. All files were used with a torque-controlled endodontic motor based on the appropriate torque and rpm values specified by the manufacturer. After determining the canal length with an electronic apex locator the apical patency was checked with a #10 K hand file. During the procedure, the canal was continuously irrigated with 5.25% sodium hypochlorite. In all irrigation procedures, a 27-gauge side-vented irrigation needle was used, which was set to be 2 mm shorter than the working length. No solvent was used during the NSER protocol. The literature has found that there is no definite consensus on the final apical diameter of the root canal when applying NSER. However, it has been reported that in primary endodontic treatment, the preparation should be completed with a larger file than the file used for apical region preparation. In this study, the final preparation was completed by using a case-specific file that was chosen to be larger than the apically compressed file while making the final preparation. The root canal was prepared with rotary files. For the final irrigation procedure is 2 mL of 5.25% NAOCl, distilled water, 17% ethylene diamine tetraacetic acid , distilled water, 2% chlorhexidine solutions were used respectively. The root canal were dried with paper points . Then, all teeth were randomly assigned one of the three study groups by using online software (http://www.random.org). (n:21).

Cold Lateral Compaction (CLC-Control Group): After the root canal preparation was completed, the working length was checked with the master cone and periapical radiography. The master cone was then covered with root canal sealer and placed in the root canal. Then, a gap was created for the .02 angled lateral cones using #30, 25 and 20 finger spreader. The obturation process continued until the spreader went 2 mm beyond the level of the canal orifice. Next, a hot excavator removed the coronal gutta-percha 1 mm below the canal orifice.

Continuous Wave Compaction (CWC): After the root canal preparation was completed, the working length was checked with the master cone and periapical radiography. Root canal sealer was applied to the root canal walls using a master cone. The plugger connected to the down-pack unit was adjusted to be 4 mm shorter than the working length. The master cone was cut 1 mm shorter than the working length with a heated plugger and applied to the root canal. Then, the heated plugger was advanced in the apical direction and the apical region was obturated. Obturation was completed in 2 stages with gutta-percha in the cartridge connected to the remaining root canal cavity back-fill unit and heated to 200 °C. Heated gutta-percha was vertically condensed with plugger to 1 in the first stage and 2 in the second. The root canal obturation was completed by removing the gutta-percha 1 mm below the canal orifice.

Thermoplasticized Gutta-Cor (TGC): After the root canal preparation was completed, the working length was controlled with the master cone and periapical radiography. Root canal sealer was applied to the root canal walls using a master cone. Root canal obturation was completed with gutta-percha heated according to the manufacturer's instructions using. The heated gutta-percha was slowly inserted into the canal up to the working length. After cutting the handle of the obturators at the level of the canal orifice with a hot excavator, it was condensed into the canal using a gutta-percha plugger. The coronal gutta-percha were removed 1 mm below the canal orifice using a hot excavator.

In the same visit, all teeth were permanently restored using direct composite resin .

ELIGIBILITY:
Inclusion Criteria

* Teeth with previously endodontic treatment but unsuccessful and developing AP, root canal obturation 2 mm shorter than the working length and teeth that do not show adequate obturation,
* Teeth with periapical lesion size less than 5mm,
* Patient with the ages of 18-65,
* Patient with dose not have systemic disease, does not use antihypertensive and antidiabetic drugs, does not have a pregnancy condition, does not use corticosteroids or antibiotics, mishaps
* Patient with no acute pain or extraoral swelling,
* Patient with no sinus tract and acute apical abscess,
* Patients with who volunteered to participate in the study and agreed to attend the control visits were included.

Exclusion Criteria

* Teeth with internal or external root resorption,
* Teeth with vertical root fracture or open apex,
* Teeth with periapical lesion size more than 5 mm,
* Patient with systemic disease,
* Patient with systemic disorders related to bone metabolism and using drugs that may affect bone metabolism,
* Patient with acute pain and therefore using analgesic medication in the last 24 hours,
* Patient with using antibiotics 2 weeks before the treatment,
* Patients who could not attend control sessions were excluded from the study .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of postoperative pain that may occur due to treatment | 1 week
  In this study, postoperative pain observed after treatment was measured using the Numeric Rating Scale (NRS).
Radiographic evaluation of healing of periapical tissues at 6 months after treatment | 6 months
  In this study, periapical radiographs obtained using a parallel film holder before and after treatment of the patients included in the study were evaluated according to the Periapical Index (PAI) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Isik M, Aydin ZU. Effect of different obturation techniques on treatment results in single-visit non-surgical endodontic retreatment: randomized controlled clinical study. BMC Oral Health. 2024 Nov 28;24(1):1449. doi: 10.1186/s12903-024-05240-3. PMID 39609817